CLINICAL TRIAL: NCT05635942
Title: Prospective Randomized Trial: Comparison Between Optimized-dose Amoxicillin and Standard-dose Amoxicillin for Quadruple Therapy in the Treatment of Helicobacter Pylori Infection in Tunisian Patients
Brief Title: Optimized-dose Amoxicillin Versus Standard-dose Amoxicillin for Quadruple Therapy in Helicobacter Pylori Eradication
Acronym: Helicomatri
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HELICO_TEST_2019
Record Dates: First submitted 2022-11-10; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori
Keywords: Disease Eradication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Technicians, who performed culture, antimicrobial susceptibility testing or urea breath test were blinded to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimized quadruple therapy (Qo-14) (Experimental): patients allocated to experimental group receive an optimized quadruple therapy (Qo-14) including 3 grams of Amoxicillin plus standard dose of clarithromycin, metronidazole and esomeprazole for 14 days.
  Interventions: Drug: optimized quadruple therapy
- standard quadruple therapy (Qs-14) (Active Comparator): patients allocated to this group receive standard quadruple therapy (Qs-14) including : amoxicillin 1g twice daily ,clarithromycin 500mg twice daily ,metronidazole 500mg twice daily and esomeprazole 40 mg twice daily for 14 days
  Interventions: Drug: standard quadruple therapy

INTERVENTIONS:
Drug: optimized quadruple therapy — Association of amoxicillin 3 g/day + Esomeprazole, nitroimidazole and clarithromycin for 14 days
  Other Names: Qo-14
  Arms: optimized quadruple therapy (Qo-14)
Drug: standard quadruple therapy — Association of amoxicillin 2 g/day + Esomeprazole, nitroimidazole and clarithromycin for 14 days
  Other Names: Qs-14
  Arms: standard quadruple therapy (Qs-14)

SUMMARY:
The goal of this prospective randomized clinical trial is to compare the rate of Helicobacter Pylori (HP) eradication after standard or dose-optimized amoxicillin quadritherapy in patients naïve to any anti-HP treatment and with chronic HP infection documented by histological examination. The main questions it aims to answer are:

* compare the eradication rate of H.Pylori after a standard concomitant quadritherapy with 2g of amoxicillin versus an optimized quadritherapy with 3g of amoxicillin, in Tunisian population
* Identify different factors associated with poor therapeutic response Patients were randomly assigned to either standard quadruple therapy (Qs-14: amoxicillin 1g twice daily, clarithromycin 500mg twice daily, metronidazole 500mg twice daily and esomeprazole 40mg twice daily for 14 days), or optimized quadruple therapy (Qo-14: amoxicillin 1g three times a day, clarithromycin 500mg twice daily, metronidazole 500mg twice daily and esomeprazole 40mg twice daily for 14 days). Eradication control was performed by urea breath test.

DETAILED DESCRIPTION:
This study was a prospective, randomized, single-center study conducted in the hepato-gastroenterology department of Mahmoud Matri Hospital in Ariana, in collaboration with the bacteriology and biochemistry laboratory of the same hospital, the anatomopathology department of Abderrahmen Mami Hospital in Ariana, and the private clinical analysis laboratory "Fendri". all patients aged from 18 and 65 years-old with H. pylori infection documented by pathological examination of per endoscopic gastric biopsies were recruited.

This was a population of patients who had undergone upper endoscopy (UE) and in whom the search for H.Pylori was indicated, according to the European Maastrich IV recommendations.

Eligible subjects were randomly assigned in a 1:1 ratio to receive either standard quadruple therapy (Qs-14) including : amoxicillin 1g twice daily ,clarithromycin 500mg twice daily ,metronidazole 500mg twice daily and esomeprazole (Medis Pharmaceutical Company) 40 mg twice daily for 14 days, or optimized quadruple therapy (Qo-14) including : amoxicillin 1g three times daily ,clarithromycin 500mg twice daily, metronidazole 500mg twice daily and esomeprazole 40 mg twice daily (Medis Pharmaceutical Company) for 14 days.

Eradication control was performed by 13C-UBT at least 4 weeks after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infection documented by pathological examination of per endoscopic gastric biopsies.

Exclusion Criteria:

* Previously received H.Pylori eradication therapy. Known allergy to one of the components of the kit used (Helikit) for 13C-urea breath test (UBT).
* A contraindication to 13C-UBT. Allergy or contraindication to the following antibiotics: Amoxicillin, Clarithromycin, Metronidazole and quinolones.
* Received antibiotics during the four weeks, or proton pump inhibitors (PPIs) during the two weeks prior to inclusion in the study.
* A history of bariatric surgery. Active gastro intestinal bleeding.
* Severe comorbidity such as decompensated cirrhosis, end-stage renal disease, decompensated cardiac disease and neoplastic disease.
* Patients on long-term immunosuppressive or corticosteroid therapy at a dose greater than 20mg/day.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
HP eeradication rate | 6 weeks after treatment completion
  Urea Breath test (UBT) is performed no sooner than 6 weeks after completion of H pylori therapy. Use of PPIs should be discontinued for at least 2 weeks before administration of the UBT.

SECONDARY OUTCOMES:
prevalence of adverse reactions | 6 weeks after treatment completion
  The percentage of patients reporting side effects during treatment and the following days until the evaluation of Hp eradication

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Kallel, PhD, Principal Investigator — Hospital Mahmoud El Matri
Locations (1):
- Hepatogastroenterology department of Mahmoud Matri Hospital, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.